CLINICAL TRIAL: NCT04815330
Title: Patient Dyspnea Under Veno-arterial Extracorporeal Circulation: Quality, Mechanisms and Sensitivity to Increased Sweep Gas Flow Through the Membrane Lung and Positive Expiratory Pressure
Brief Title: Patient Dyspnea Under Veno-arterial Extracorporeal Circulation
Acronym: DYSCO2
Status: Completed | Type: Observational
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00539-30
Record Dates: First submitted 2021-02-10; First posted 2021-03-25 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Dyspnea
Keywords: Patient-ventilator interaction; Veno-arterial extracorporeal circulation; Inspiratory muscles; Electromyogram; Mechanical ventilation
MeSH Terms: conditions — Dyspnea | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient dyspnea under veno-arterial extracorporeal circulation: Relief of dyspnea will be carried out by the clinician in charge of the patient. He will have complete control of his behaviour. He will carry out this test according to the practices in force in the department.
  If a sweep gas flow through the membrane lung increment has been decided upon to relieve dyspnea, a new recording will be made after each scan increment and the patient will be asked at each step.
  In ventilated or non-ventilated patients in whom the decision to implement non-invasive ventilation has been made, an increase in PEEP in 2 cmH2O steps without exceeding a plateau pressure of 25 cmH2O and a VT of 10ml/kg of the patient's theoretical weight will be achieved.
  Interventions: Other: increment sweep gas flow; Other: non-invasive ventilation

INTERVENTIONS:
Other: increment sweep gas flow — If a sweep gas flow through the membrane lung increment has been decided upon to relieve dyspnea, a new recording will be made after each scan increment and the patient will be asked at each step.
Other: non-invasive ventilation — In ventilated or non-ventilated patients in whom the decision to implement non-invasive ventilation has been made, an increase in PEEP in 2 cmH2O steps without exceeding a plateau pressure of 25 cmH2O and a VT of 10ml/kg of the patient's theoretical weight will be achieved.

SUMMARY:
Rationale: Patients with severe heart failure increasingly benefit from extracorporeal circulatory assistance (Extracorporeal Membrane Oxygenation - ECMO) that completely replaces the function of the heart and is in addition to mechanical ventilation (veno-arterial ECMO). In clinical practice, some of these patients have been found to be dyspneic, although circulatory assistance ensures satisfactory hematosis. Indeed, nearly half of the patients undergoing mechanical ventilation in intensive care have a generally intense dyspnea. In addition to the immediate discomfort caused by dyspnea, which can be assimilated to pain, this symptom is associated with a prolonged duration of mechanical ventilation and contributes to the genesis of neuropsychological sequelae of resuscitation such as post-traumatic stress syndrome.

Objectives :

1. To study the effectiveness and impact of an increase in ECMO sweep gas flow through the membrane lung or positive tele-expiratory pressure (PEP) on dyspnea in patients under ECMO.
2. To understand the mechanism involved in this relief of dyspnea. Methods: in 30 patients of Intensive Care Unit, dyspnea will be evaluated by psychophysiological scales and scores as well as by neurophysiological tools (electromyography of inspiratory muscles) during sweep gas flow through the membrane lung incrementation and PEP increase.

Ethical framework: Changes in ventilation parameters and ECMO will be performed in the usual manner, without additional or unusual diagnostic, treatment or monitoring procedures.

Expected results and outlook: the investigators hypothesize that half of the patients on veno-arterial ECMO have dyspnea related to pulmonary edema. Therefore, an increase in PEP would alleviate this dyspnea. The investigators hypothesize that by using a relief method related to increased sweep gas flow through the membrane lung, the investigators can reduce the discomfort without inducing any associated complication.

This study will improve the knowledge of the mechanisms determining dyspnea in patients under ECMO and the principle of therapeutic strategy to improve it.

DETAILED DESCRIPTION:
Half of the patients undergoing mechanical ventilation in intensive care have moderate to severe dyspnea. This dyspnea has a negative impact on the prognosis and quality of life in the medium term.

As ECMOs, techniques for extracorporeal assistance to supplement cardiac and pulmonary functions, are developing rapidly, it seems essential to study the dyspnea associated with the use of these techniques. In particular, understanding the main mechanisms involved in the genesis of dyspnea in patients under ECMO would allow the development of therapeutic solutions aimed at minimizing it.

The investigators hypothesize that, in patients under veno-arterial ECMO with dyspnea, the dyspnea decreases in response to an increase in ECMO sweep gas flow through the membrane lung via modulation of central and peripheral chemoreceptors sensitive to variations in PaO2, PaCO2 and pH. Since dyspnea experienced by patients on veno-arterial ECMO is related to cardiogenic pulmonary edema, increased discharge from the left cavities by increasing positive expiratory pressure should also alleviate dyspnea.

The main objective of the present study is to evaluate the impact of sweep gas flow through the membrane lung and PEP incrementation on dyspnea in patients with veno-arterial ECMO with dyspnea.

Relief of dyspnea will be carried out by the clinician in charge of the patient. He will have complete control of his behaviour. He will carry out this test according to the practices in force in the department.

One of the investigators will be present and will collect the data listed above. This investigator will not intervene in the conduct of the test.

Each patient will participate in a dyspnea relief test according to the protocol of the department and according to the management of the practitioner in charge of the patient.

Initially a recording of 5 minutes will be made in the basal state, before any therapeutic action.

If a sweep gas flow through the membrane lung increment has been decided upon to relieve dyspnea, a new recording will be made after each scan increment and the patient will be asked at each step.

In ventilated or non-ventilated patients in whom the decision to implement non-invasive ventilation has been made, an increase in PEEP in 2 cmH2O steps without exceeding a plateau pressure of 25 cmH2O and a VT of 10ml/kg of the patient's theoretical weight will be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Circulatory support by veno-arterial ECMO for cardiogenic shock;
* Presence of severe respiratory distress;
* Presence of dyspnea ≥ 40 mm on a visual analogue scale of dyspnea (VAS-dyspnea)
* Decision by the clinician in charge of the patient to either modify the ECMO parameters or to administer non-invasive ventilation in order to decrease the intensity of the dyspnea;
* presence of an arterial catheter; :
* RASS score between 0 and +1 ;
* Absence of delirium on the CAM-ICU score;
* being socially insured.

Exclusion Criteria:

* patient unable to express opposition;
* protected minor or adult patient;
* pregnant woman;
* double veno-arterial ECMO; central ECMO; left ventricular assist or long-term bi-ventricular assist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under veno-arterial ECMO with dyspnea
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Dyspnea change | Baseline, during the intervention
  A quantification of dyspnea will be carried out by visual analogue dyspnea scale (D-VAS). This scale with a cursor will be presented vertically to the patient at inclusion, then at the end of each period and will be graduated from 0 (no dyspnea) to 100 (maximum dyspnea). The patient will indicate the intensity of the dyspnea with a slider;

SECONDARY OUTCOMES:
Arterial Blood Gas | Baseline, during the intervention
  If an arterial blood gas measurement is performed at the clinician's request, the results will be collated.
Electromyogram (EMG) of extra-diaphragmatic inspiratory muscles | Baseline, during the intervention
  The amplitude of the EMG signal of the extra-diaphragmatic inspiratory muscles is proportional to the intensity of the dyspnea. The EMG will be collected by self-adhesive surface electrodes of the same type as those usually used to collect the ECG signal in ICU patients. A distance of 2 cm will separate the two electrodes. The impedance should be less than 2000 Ω. The position of the electrodes will depend on the muscle whose EMG activity is being collected:
  * parasternal intercostal muscles: opposite the 2nd intercostal space, as close as possible to the sternum;
  * Alae nasi muscles: on the wings of the nose.
Evaluation of pain | Baseline, during the intervention
  Pain: Pain will be assessed using a visual analog scale ranging from 0 ("no pain") to 100 ("maximum pain").

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Demoule, MD, PhD, Principal Investigator — Groupe Hospitalier Universitaire APHP - Sorbonne Université Site Pitié-Salpêtrière (bâtiment Eole)
Locations (1):
- Service de Pneumologie et Réanimation Médicale, Groupe Hospitalier Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No